CLINICAL TRIAL: NCT06939582
Title: A Single Center, Open Label Phase II Clinical Trial of Hydroxychloroquine Sulfate Tablets for the Treatment of Radiation Stomatitis and Taste Disturbance in Intensity Modulated Radiotherapy for Head and Neck Cancer
Brief Title: Hydroxychloroquine Sulfate Tablets for Radiation-induced Oral Mucositis
Acronym: RIOM
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Xingchen Peng (Other)
Responsible Party: Sponsor-Investigator, Xingchen Peng, Department of Radiation Oncology, Clinical Professor，West China Hospital, West China Hospital
Organization: West China Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20241413
Record Dates: First submitted 2025-04-20; First posted 2025-04-23 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Radiation-induced Oral Mucositis
MeSH Terms: interventions — Hydroxychloroquine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control group (Placebo Comparator): use the placebo
  Interventions: Other: Placebo
- trial group (Experimental): use the hydroxychloroquine sulfate tablets
  Interventions: Drug: Hydroxychloroquine Sulfate Tablets

INTERVENTIONS:
Drug: Hydroxychloroquine Sulfate Tablets — the trial group use the hydroxychloroquine sulfate tablets (200mg/time, bid)
  Arms: trial group
Other: Placebo — the control group use the Placebo
  Arms: Control group

SUMMARY:
Evaluate the safety, tolerance and efficacy of hydroxychloroquine sulfate tablets the prevention and treatment of oral mucositis and dysgeusia in patients undergoing radiotherapy

ELIGIBILITY:
Inclusion Criteria:

* Patients pathologically diagnosed with non-metastatic head and neck malignant tumors
* Aged 18-80 years
* Eastern Cooperative Oncology Group performance status of ≤2
* Planning to receive definitive RT or postoperative adjuvant RT
* Normal liver, kidney and bone marrow function
* Sign informed consent

Exclusion Criteria:

* Those who are known to be allergic to 4-aminoquinoline compounds or have more serious allergic constitution
* Had a history of head and neck radiotherapy
* Patients with non head and neck parts in the radiotherapy area
* Poor oral hygiene or severe periodontitis
* Suffering from severe kidney disease, severe cardiovascular disease, myasthenia gravis, Parkinson's disease or epilepsy
* Recently taking or taking diuretics or other drugs known to interact with hydroxychloroquine sulfate tablets
* Retinopathy
* Other patients (combined with any serious other diseases) who the investigator believes are not suitable for participation in this study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 158 (Estimated)
Dates: Start 2024-12-22 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-06-20 (Estimated)

PRIMARY OUTCOMES:
the WHO grade of RIOM | From the start of radiotherapy to 8 weeks after completion of radiotherapy
  use the WHO Oral Toxicity Scale to evaluate the WHO grade of RIOM. WHO O grade: no representation of RIOM; WHO 1 grade: soreness and erythema; WHO 2 grade: erythema, ulcers and ability to eat solids; WHO 3 grade: ulcers, requiring liquid diet; WHO 4 grade: alimentation not possible. The higher scores mean a worse outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Radiation Oncology, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Schrezenmeier E, Dorner T. Mechanisms of action of hydroxychloroquine and chloroquine: implications for rheumatology. Nat Rev Rheumatol. 2020 Mar;16(3):155-166. doi: 10.1038/s41584-020-0372-x. Epub 2020 Feb 7. PMID 32034323